CLINICAL TRIAL: NCT04314583
Title: Feasibility of a Gratitude Intervention for Cardiac Rehabilitation Patients: A Nursing-based Intervention
Brief Title: Gratitude Intervention for Cardiac Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martha Biddle (Other)
Responsible Party: Sponsor-Investigator, Martha Biddle, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 57514
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases
Keywords: depression; pessimism; gratitude; nursing
MeSH Terms: conditions — Cardiovascular Diseases; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control Group (Active Comparator): Adult patients attending cardiovascular rehabilitation.
  Interventions: Behavioral: Attention Control
- Gratitude Journaling Group (Experimental): Adult patients attending cardiovascular rehabilitation.
  Interventions: Behavioral: Gratitude Journaling

INTERVENTIONS:
Behavioral: Attention Control — Participants in this group will be asked to recall 3 to 5 events from the prior day of the intervention and write, or if unable to write, speak about these events.
  Arms: Attention Control Group
Behavioral: Gratitude Journaling — The gratitude journaling intervention involves participants writing or speaking 3-5 things for which they are grateful and focusing on these attributes. Participants will do this weekly for 12 weeks.
  Arms: Gratitude Journaling Group

SUMMARY:
This is a single-center cohort study of patients in a cardiac rehabilitation program with a diagnosis of cardiovascular disease (CVD), including heart failure, coronary artery disease, post myocardial infarction, post percutaneous coronary intervention and post cardiac surgery. Participants will be randomized to the gratitude intervention or an attention control group. This study is a pilot study to determine the feasibility and acceptability of administering the gratitude intervention in a cardiac rehabilitation setting.

DETAILED DESCRIPTION:
Nursing-led interventions of chronic diseases, including cardiovascular disease (CVD), have been proved to be successful. Appropriately trained nurses produce high-quality care and good health outcomes for patients equivalent to that achieved by physicians with higher levels of patient satisfaction. CVD, including coronary artery disease and heart failure, is a major and rapidly growing public health problem. Despite advances in its treatment, it remains the leading cause of death in the U.S. Furthermore, the prevalence of CVD in adults is estimated to continue to rise and that by 2035, 45.1% of the U.S. population will have some form of CVD with total costs expected to reach $1.1 trillion with direct medical costs projects to reach $748.7 billion. Therefore, novel preventive efforts are needed.

Negative psychological states, including depression and pessimism (negative future expectation), have been linked with poor CVD outcomes. Despite the fact that optimism (positive future expectation) and other positive affective states have been associated with superior cardiovascular outcomes, little research has focused on interventions designed to increase positive psychological states in patients at risk for CVD. In the current trial, patients in an academic medical center cardiac rehabilitation program will be approached. Cardiac rehabilitation is an integral component in the treatment of patients with cardiovascular disease including coronary artery disease, heart failure with reduced ejection fraction, following heart valve surgery or cardiac transplantation.

One of its core components is psychological support and management. In this nursing-led study, participants will be randomized to a gratitude intervention or an attention control group. The gratitude intervention, which encourages participants to notice and appreciate the positive features of life, is based on the work of Emmons and McCullough, and involves participants writing (or if unable to write, speaking) things for which they are grateful. Much of the existing research on gratitude (noticing and appreciating the positive features of life) has focused primarily on outcomes associated with psychological factors and social interactions.

The primary aim of this feasibility study will be to determine if a gratitude intervention is acceptable and feasible in a cohort of patients attending cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* able to consent
* patient at cardiac rehabilitation program at Gill Heart and Vascular Institute

Exclusion Criteria:

- under the age of 18

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Percent Completion of Cardiac Rehabilitation Program | 12 weeks
  Percentage of patients in each arm who complete the cardiac rehabilitation program.

SECONDARY OUTCOMES:
Change in Gratitude | 12 weeks
  The Gratitude Questionaire (GQ6) will be used to assess gratitude at baseline and following the intervention. The GQ6 is a 6 item questionnaire with scales ranging from 1-7. Cumulative scores range from 6-42; higher scores indicate increased gratitude.
Change in Dispositional Optimism | 12 weeks
  The Life Orientation Test-Revised (LOT-R) will be used to assess optimism at baseline and following the intervention. The LOT-R is a 10-item survey, with scales ranging from 1-5. (Not all questions are scored). Cumulative scores range from 6-30; higher scores indicate increased optimism.
Change in Resilience | 12 weeks
  The Brief Resilience Scale (BRS) will be used to measure resilience at baseline and after the intervention. The BRS is a 6 item survey, with each item scored from 1-5. Raw total scores range from 6-30; final scores will be calculated as the mean of all scores. Higher scores indicate increased resiliency.
Hospital Readmission | one year
  Percent of patients readmitted to the hospital
Mortality | one year
  Percent of patients deceased

CONTACTS AND LOCATIONS:
Overall Officials: Martha Biddle, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No